CLINICAL TRIAL: NCT01587716
Title: A Randomised, Double-blind, Placebo Controlled, Inhaled Single Escalating and Repeat Dose Study Using an Aqueous Droplet Inhaler to Investigate the Safety, Tolerability and Pharmacokinetics of GSK2339345.
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK2339345.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115658
Record Dates: First submitted 2012-04-19; First posted 2012-04-30 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Cough
Keywords: Safety and tolerability, pharmacokinetics, cough, voltage gated sodium channels (VGSC), anaesthesia
MeSH Terms: conditions — Cough | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1. Inhaled GSK2339345/Placebo Single Dose (Cohort 1) (Experimental): administered three ascending doses of GSK2339345 or placebo as a solution via an aqueous droplet inhaler over four treatment periods, with at least 5 days washout between doses
  Interventions: Drug: GSK2339345 (Inhaled) Single Dose; Other: Placebo (Inhaled) Single Dose
- 2. Inhaled GSK2339345/Placebo Repeat Dose (Cohort 2) (Experimental): administered a dose of GSK2339345 or placebo, four times a day on two consecutive days. Each subject will receive either GSK2339345 or matching placebo as a solution administered via an aqueous droplet inhaler
  Interventions: Drug: GSK2339345 (Inhaled) Repeat Dose; Other: Placebo (Inhaled) Repeat Dose

INTERVENTIONS:
Drug: GSK2339345 (Inhaled) Single Dose — 250, 1000 and 2000 microgram (proposed doses)
  Arms: 1. Inhaled GSK2339345/Placebo Single Dose (Cohort 1)
Other: Placebo (Inhaled) Single Dose — Inhaled 0.9% sodium chloride solution
  Arms: 1. Inhaled GSK2339345/Placebo Single Dose (Cohort 1)
Drug: GSK2339345 (Inhaled) Repeat Dose — 2000 microgram (proposed dose) administered 4 times a day for two consecutive days
  Arms: 2. Inhaled GSK2339345/Placebo Repeat Dose (Cohort 2)
Other: Placebo (Inhaled) Repeat Dose — Inhaled 0.9% sodium cholride solution
  Arms: 2. Inhaled GSK2339345/Placebo Repeat Dose (Cohort 2)

SUMMARY:
This is a study of the sodium channel inhibitor, GSK2339345. Cohort 1 will assess the safety, tolerability and PK of single ascending doses of GSK2339345 administered via an aqueous droplet inhaler in healthy subjects. Cohort 2 will assess the safety, tolerability, and PK of repeat doses of GSK2339345 administered four times a day for two consecutive days via an aqueous droplet inhaler.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics (PK) effects of GSK2339345 in healthy subjects. GSK2339345 is a blocker of neuronal voltage gated sodium channels in development for the treatment of chronic cough, excessive cough and post-viral and viral (acute) cough. Inhaled pan NaV inhibitors are associated with oropharyngeal sensation perturbation and so this study will establish the potential local sensate effects of GSK2339345 at multiples of the predicted inhaled therapeutic dose. This study also aims to define the maximum tolerated dose of GSK2339345 administered via an aqueous droplet inhaler. Cohort 1 is a randomised, double-blind, placebo-controlled, cross-over, inhaled single-dose escalating study using an aqueous droplet inhaler. Cohort 1 will include assessments of sensate changes via a 4 point scale, assessment of taste via an 11 point scale, and PK assessments to investigate the PK profile of GSK2339345. Cohort 2 of this study is a randomised, double blind, placebo controlled, parallel group, inhaled repeat dose study using a aqueous droplet inhaler. Subjects will be randomised to receive 2000 microgram of GSK2339345 or placebo four times a day for two consecutive study days. Similar assessments of sensations to those used in Cohort 1 will be performed. The potential for systemic cardiovascular (CV) or central nervous system (CNS) effects will also be assessed throughout the study via observation. Cohort 2 will also include PK assessments to investigate the PK profile of GSK2339345. Placebo will be used throughout the study as a control.

ELIGIBILITY:
Inclusion Criteria:

* ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Average QTcB < 450 msec
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Non-smoker for at least 6 months with a pack history ≤ 5pack years (Pack years = (No. of cigarettes smoked/day/20) x No. of years smoked).
* Body weight ≥ 50 kg and BMI within the range 19 - 32.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* A 24 hour Holter ECG at screening that demonstrates no clinically significant abnormalities or finding that could interfere with interpretation of the study results, when assessed by an appropriately trained and experienced reviewer.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Current or chronic history of cardiovascular disease (e.g. hypertension, coronary heart disease, heart attack, angina, myocardial infarct, and stroke).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

  • An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* FEV1 less than 80% of the predicted value prior to dosing.
* Any subject who, upon oropharyngeal examination, is deemed by the Investigator to be unsuitable for oropharyngeal sensation assessments. This includes any injuries to the mucosa of the mouth or pharynx that could potentially increase systemic absorption e.g candidiasis.
* Any subject who has a history of an allergic reaction to a local anaesthetic. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Subjects who have asthma or a history of asthma.
* Breath CO levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Subjects who are unable to use the inhaler satisfactorily.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04-23 (Actual); Primary Completion 2012-07-30 (Actual); Study Completion 2012-07-30 (Actual)

PRIMARY OUTCOMES:
Safety parameters: AEs, vital signs, ECG, body temperature and laboratory assessments, including haematology, clinical biochemistry and cardiac troponin. | Approximately 5 weeks from first dose to the follow-up visit.
  To assess the safety and tolerability of single and repeat inhaled doses of GSK2339345 administered by an aqueous droplet inhaler.
Assessment of oropharyngeal sensation perturbation via a 4 point scale. | Approximately 5 weeks from first dose to the follow-up visit.
  To assess the changes in oropharyngeal sensation caused by single and repeat inhaled doses of GSK2339345 administered by an aqueous droplet inhaler.

SECONDARY OUTCOMES:
Plasma concentrations of GSK2339345 and single and repeat dose derived pharmacokinetic parameters including Cmax, tmax, AUC(0-t), AUC(0-inf), and AUC(0- τ), as appropriate where data allow. | Approximately 5 weeks from first dose to the follow-up visit.
  To evaluate the systemic pharmacokinetics of single and repeat doses of inhaled GSK2339345 in healthy volunteers administered by an aqueous droplet inhaler.
Identification of taste of the solution and rating on 11 point scale to rate pleasantness or unpleasantness | Approximately 5 weeks from first dose to the follow-up visit.
  To assess the palatability of GSK2339345 administered by an aqueous droplet inhaler

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115658 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115658?search=study&search_terms=115658#rs
- Available data/document: Dataset Specification: 115658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115658 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register